CLINICAL TRIAL: NCT05055414
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel, Phase 2 Study to Evaluate the Efficacy and Safety of UI030 in COVID-19 Patients
Brief Title: Arformoterol/Budesonide for COVID-19
Acronym: ABC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUP-UI030-231
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UI030 (Experimental): UI030 (Budesonide/Arformoterol dry powder inhaler, 3 inhalations b.i.d at 3 days and 2 inhalations b.i.d at 11 days) or placebo for 2 weeks.
  Interventions: Drug: UI030
- Placebo (Placebo Comparator): UI030 (Budesonide/Arformoterol dry powder inhaler, 3 inhalations b.i.d at 3 days and 2 inhalations b.i.d at 11 days) or placebo for 2 weeks.
  Interventions: Drug: UI030

INTERVENTIONS:
Drug: UI030 — Budesonide/Arformoterol dry powder inhaler, 3 inhalations b.i.d at 3 days and 2 inhalations b.i.d at 11 days

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel, phase 2 study to evaluate the efficacy and safety of UI030 in COVID-19 patients

DETAILED DESCRIPTION:
Patients with moderate and severe COVID-19 were randomly assigned (1:1) to receive either UI030 (Budesonide/Arformoterol dry powder inhaler, 2 inhalations b.i.d) or placebo for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult, aged 19 years or above
* New onset of symptoms suggestive of COVID-19 (fever, cough, soar throat, etc) or diagnosed with COVID-19 within 7 days of participant being seen at visit 1
* In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

* A condition requiring invasive oxygen support;
* History of hypersensitivity to budesonide and arformoterol
* Pregnancy, Breast-feeding
* Participation in other clinical studies within 4 weeks prior to enrollment in this study.
* Refusal of the patient to continue participating in the study/withdrawal of informed consent by the patient.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Improvement on World Health Organization (WHO) Ordinal Scale | 28 days
  The median time to reach the clinical improvement on the WHO Ordinal 9 Scale for Clinical Improvement [0-8]

SECONDARY OUTCOMES:
World Health Organization (WHO) Ordinal Scale for Clinical Improvement | 28 days
  Improvement rate of patients with WHO Clinical Ordinal 9 Scale [0-8]
World Health Organization (WHO) Ordinal Scale change | 28 days
  Change from baseline in WHO Ordinal 9 Scale [0-8]
Clinical cure rate | 28 days
  Percentage of patients with clinical cure and improvement